CLINICAL TRIAL: NCT03924791
Title: Transforaminal Epidural Injection in Acute Sciatica
Acronym: TEIAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C.L.A.Vleggeert-Lankamp (Other)
Collaborators: Spaarne Gasthuis (Other); Stichting Achmea Gezondheidszor (Other); Posthumus Meyjes Fonds (Unknown)
Responsible Party: Sponsor-Investigator, C.L.A.Vleggeert-Lankamp, Dr. C.L.A. Vleggeert-Lankamp, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEIAS
Record Dates: First submitted 2019-04-10; First posted 2019-04-23 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Sciatica; Sciatica Due to Intervertebral Disc Disorder; Sciatic Radiculopathy
Keywords: Sciatica; Acute sciatica; Transforaminal epidural injection; Leg pain; Lumbar spine; Back pain; Lumbar surgery; Herniated intervertebral lumbar disk; Cost-effectiveness
MeSH Terms: conditions — Sciatica; Back Pain | interventions — Lidocaine; Methylprednisolone Acetate; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either treatment with transforaminal epidural injection or standard oral pain medication.
Masking Description: Since masking is not possible for treatment with injections and oral pain medication, this is an open-label study. Outcomes are assessed by patients through online questionnaires and therefore the outcome assessor is not masked as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transforaminal Epidural Injection (Experimental): Transforaminal Epidural Injection containing 1,5 mL lidocaine 2% and 40mg methylprednisolone acetate for injections L3 or below Transforaminal Epidural Injection containing 1,5 mL lidocaine 1% and 10mg dexamethasone for injections above L3
  Interventions: Drug: Lidocaine; Drug: Methylprednisolone Acetate; Drug: Dexamethasone
- Oral pain medication (No Intervention): Patients will receive oral pain medication according to general practitioner guidelines.

INTERVENTIONS:
Drug: Lidocaine — In combination with dexamethasone or methylprednisolone acetate
  Arms: Transforaminal Epidural Injection
Drug: Methylprednisolone Acetate — In combination with lidocaine
  Other Names: Depo-Medrol
  Arms: Transforaminal Epidural Injection
Drug: Dexamethasone — In combination with lidocaine
  Arms: Transforaminal Epidural Injection

SUMMARY:
Patients suffering from sciatica are treated conservatively for the first 8 weeks due to the favourable prognosis. This period is preferably extended up to 14-16 weeks after which patients may opt for surgery. However, patients may experience severe discomfort due to pain in the leg which can lead to decreased physical activity and socio-economic problems. An adequate therapy to alleviate symptoms during this period of 'wait-and-see' is lacking. In this study, patients will be randomized to treatment with transforaminal epidural injections or standard oral pain medication.

DETAILED DESCRIPTION:
Sciatica is a condition of radicular pain in the leg and is usually caused by herniation of a lumbar intervertebral disc. The herniated disc compresses a lumbar nerve root that continues its route into the sciatic nerve. About 13% to 40% of all people will suffer from sciatica at least once during their lifetime. Sciatica can have severe socio-economic effects; patients are immobilised by the pain they experience and therefore cannot go to work or participate in social events. Most cases resolve spontaneously with conservative therapy using only standard analgesics and/or physiotherapy. In a large RCT it was demonstrated that outcome of conservative and surgical therapy was comparable after 26 weeks. With this knowledge the guidelines for surgical treatment of sciatica were adjusted and it is nowadays usual care to offer surgery only after at least 8 weeks of conservative care and preferably after 14-16 weeks of conservative care. This decision is made together with the patient in a process of Shared Decision making. Although this treatment regimen has been demonstrated to be efficacious and cost effective, the burden for a patient during these weeks of conservative care is usually high. The investigators seek to find a type of conservative care to reduce the discomfort due to the pain and to enable the patient to remain physically active. Not only will this add to the quality of life of the patient, but it will also prevent the patient from taking a sick-leave. In this study, patients will be randomized to either treatment with transforaminal epidural injections or to standard care consisting of oral pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sciatica by GP
* NRS leg pain of 6 or more on a 10-point NRS scale
* Minimum duration of symptoms of 3 weeks and maximum duration of 8 weeks

Exclusion Criteria:

* Age under 18 years
* Condition preventing to receive transforaminal epidural injection
* Severe scoliosis
* Transforaminal epidural injection received in 6 months before randomization date
* Surgery for sciatica at the same level
* Surgery for sciatica at another level within one year before inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) for leg pain | 2 weeks after randomization
  Pain intensity in the leg using the NRS. 0 is the minimal score indicating no pain, 10 is the maximum indicating the worst imaginable pain. Scale increases with increments of 1.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for leg pain | Baseline, 1, 4, 10 and 21 weeks after randomization
  Pain intensity in the leg using the NRS. 0 is the minimal score indicating no pain, 10 is the maximum indicating the worst imaginable pain. Scale increases with increments of 1.
Numerical Rating Scale (NRS) for back pain | Baseline, 1, 2, 4, 10 and 21 weeks after randomization
  Pain intensity in the back using the NRS. 0 is the minimal score indicating no pain, 10 is the maximum indicating the worst imaginable pain. Scale increases with increments of 1.
Oswestry Disability Index (ODI) | Baseline, 1, 2, 4, 10 and 21 weeks after randomization
  Assessment of functionality using the ODI. 0 is the minimal score indicating no disability, 50 is the maximum indicating the worst disability possible. This questionnaire is based on 10 questions with answers corresponding to values of 0-5 points.
EuroQoL Cost Utility (EQ-5D) | Baseline, 2, 10 and 21 weeks after randomization
  Assessment of cost utility using the EuroQoL EQ-5D analysis tool. The tool measures five dimensions: mobility, self-care, daily activities, pain/discomfort and anxiety/depression.
Quality of Life Visual Analogue Scale | Baseline, 2, 10 and 21 weeks after randomization
  Assessment of the utility by valuation of the patient's health state representing the patient's perspective. 0 is the minimal score indicating 'as bad as death', 100 is the maximum indicating 'perfect health'. Scale increases with increments of 1.
Likert scale | Baseline, 1, 2, 4, 10 and 21 weeks after randomization
  Perceived recovery by the patient using the Likert scale. This is a 7-point scoring scale that ranges from 'completely recovered' to 'worse than ever'.
Cost diary | 10 and 21 weeks after randomization
  Determination of medical expenses due to health care utilization (costs of medication, physiotherapy, treatment by a medical specialist), patient costs (mobility aid, nursing care, domestic help), and absenteeism from work (amount of hours of absenteeism, hourly wage).
Complications from treatment with transforaminal epidural injection (TEI) | Throughout the follow-up of 21 weeks
  The occurrence and incidence of complications caused by treatment with TEI will be reported.
Level and shape of disc herniation from MRI data | 21 weeks after randomization
  The lumbar intervertebral level and shape of the herniated disc will be described based on MRI data
Size of disc herniation from MRI data | 21 weeks after randomization
  The size of the herniated disc will be reported in millimetres based on MRI data
Pfirrmann scale for disc degeneration on MRI | 21 weeks after randomization
  Disc degeneration on MRI will be assessed using the Pfirrmann scale which distinguishes 5 degrees of disc degeneration. Grade 1 indicates a normal disc. Higher grades indicate a more severe degenerative state of the intervertebral disc.
Histology of disc material obtained during surgery | 21 weeks after randomization
  Identification of immunological cells, macrophages and bacteria in disk material obtained during discectomy using staining, cell culture and polymerase chain reaction techniques.
Modic scale for end plate changes on MRI | 21 weeks after randomization
  The degree of end plate changes on MRI will be assessed using the Modic scale which distinguishes 3 degrees of end plate changes. All three Modic degrees indicate a certain type of underlying pathology in the vertebra. When the vertebra is normal, Modic changes are absent.
Weishaupt scale for facet degeneration on MRI | 21 weeks after randomization
  The degree of facet degeneration on MRI will be assessed using the Weishaupt scale which distinguishes 4 degrees of facet degeneration. Grade 0 indicates normal facet joint space. Higher grades indicate a more severe degenerative state of the facet joint.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen LA Vleggeert-Lankamp, MD Msc Ph.D, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Spaarne Gasthuis, Haarlem
  - Spaarne Gasthuis, Hoofddorp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peul WC, van Houwelingen HC, van den Hout WB, Brand R, Eekhof JA, Tans JT, Thomeer RT, Koes BW; Leiden-The Hague Spine Intervention Prognostic Study Group. Surgery versus prolonged conservative treatment for sciatica. N Engl J Med. 2007 May 31;356(22):2245-56. doi: 10.1056/NEJMoa064039. PMID 17538084
- [Background] Hofstede SN, van Bodegom-Vos L, Wentink MM, Vleggeert-Lankamp CL, Vliet Vlieland TP, Marang-van de Mheen PJ; DISC study group. Most important factors for the implementation of shared decision making in sciatica care: ranking among professionals and patients. PLoS One. 2014 Apr 7;9(4):e94176. doi: 10.1371/journal.pone.0094176. eCollection 2014. PMID 24710328
- [Background] Joswig H, Neff A, Ruppert C, Hildebrandt G, Stienen MN. The Value of Short-Term Pain Relief in Predicting the Long-Term Outcome of Lumbar Transforaminal Epidural Steroid Injections. World Neurosurg. 2017 Nov;107:764-771. doi: 10.1016/j.wneu.2017.08.055. Epub 2017 Aug 23. PMID 28838872
- [Background] Spijker-Huiges A, Vermeulen K, Winters JC, van Wijhe M, van der Meer K. Epidural steroids for lumbosacral radicular syndrome compared to usual care: quality of life and cost utility in general practice. Arch Phys Med Rehabil. 2015 Mar;96(3):381-7. doi: 10.1016/j.apmr.2014.10.017. Epub 2014 Nov 8. PMID 25448243
- [Background] Kuslich SD, Ulstrom CL, Michael CJ. The tissue origin of low back pain and sciatica: a report of pain response to tissue stimulation during operations on the lumbar spine using local anesthesia. Orthop Clin North Am. 1991 Apr;22(2):181-7. PMID 1826546
- [Background] Takahashi H, Suguro T, Okazima Y, Motegi M, Okada Y, Kakiuchi T. Inflammatory cytokines in the herniated disc of the lumbar spine. Spine (Phila Pa 1976). 1996 Jan 15;21(2):218-24. doi: 10.1097/00007632-199601150-00011. PMID 8720407
- [Background] El Barzouhi A, Vleggeert-Lankamp CL, Lycklama A Nijeholt GJ, Van der Kallen BF, van den Hout WB, Verwoerd AJ, Koes BW, Peul WC; Leiden-The Hague Spine Intervention Prognostic Study Group. Magnetic resonance imaging interpretation in patients with sciatica who are potential candidates for lumbar disc surgery. PLoS One. 2013 Jul 10;8(7):e68411. doi: 10.1371/journal.pone.0068411. Print 2013. PMID 23874616
- [Background] Verwoerd AJ, Peul WC, Willemsen SP, Koes BW, Vleggeert-Lankamp CL, el Barzouhi A, Luijsterburg PA, Verhagen AP. Diagnostic accuracy of history taking to assess lumbosacral nerve root compression. Spine J. 2014 Sep 1;14(9):2028-37. doi: 10.1016/j.spinee.2013.11.049. Epub 2013 Dec 8. PMID 24325881
- [Background] el Barzouhi A, Vleggeert-Lankamp CL, Lycklama a Nijeholt GJ, Van der Kallen BF, van den Hout WB, Koes BW, Peul WC; Leiden-The Hague Spine Intervention Prognostic Study Group. Reliability of gadolinium-enhanced magnetic resonance imaging findings and their correlation with clinical outcome in patients with sciatica. Spine J. 2014 Nov 1;14(11):2598-607. doi: 10.1016/j.spinee.2014.02.028. Epub 2014 Feb 21. PMID 24561397
- [Background] el Barzouhi A, Vleggeert-Lankamp CL, Lycklama a Nijeholt GJ, Van der Kallen BF, van den Hout WB, Koes BW, Peul WC; Leiden-The Hague Spine Intervention Prognostic Study Group. Influence of low back pain and prognostic value of MRI in sciatica patients in relation to back pain. PLoS One. 2014 Mar 17;9(3):e90800. doi: 10.1371/journal.pone.0090800. eCollection 2014. PMID 24637890
- [Background] Verwoerd AJH, Mens J, El Barzouhi A, Peul WC, Koes BW, Verhagen AP. A diagnostic study in patients with sciatica establishing the importance of localization of worsening of pain during coughing, sneezing and straining to assess nerve root compression on MRI. Eur Spine J. 2016 May;25(5):1389-1392. doi: 10.1007/s00586-016-4393-8. Epub 2016 Feb 2. PMID 26842881
- [Background] El Barzouhi A, Verwoerd AJ, Peul WC, Verhagen AP, Lycklama A Nijeholt GJ, Van der Kallen BF, Koes BW, Vleggeert-Lankamp CL; Leiden-The Hague Spine Intervention Prognostic Study Group. Prognostic value of magnetic resonance imaging findings in patients with sciatica. J Neurosurg Spine. 2016 Jun;24(6):978-85. doi: 10.3171/2015.10.SPINE15858. Epub 2016 Feb 12. PMID 26871651
- [Background] Katz NP, Paillard FC, Ekman E. Determining the clinical importance of treatment benefits for interventions for painful orthopedic conditions. J Orthop Surg Res. 2015 Feb 3;10:24. doi: 10.1186/s13018-014-0144-x. PMID 25645576
- [Background] Joswig H, Neff A, Ruppert C, Hildebrandt G, Stienen MN. The Value of Short-Term Pain Relief in Predicting the One-Month Outcome of Lumbar Transforaminal Epidural Steroid Injections. World Neurosurg. 2016 Dec;96:323-333. doi: 10.1016/j.wneu.2016.09.016. Epub 2016 Sep 15. PMID 27641258
- [Derived] Verheijen E, Munts AG, van Haagen O, de Vries D, Dekkers O, van den Hout W, Vleggeert-Lankamp C. Transforaminal epidural injection versus continued conservative care in acute sciatica (TEIAS trial): study protocol for a randomized controlled trial. BMC Neurol. 2019 Sep 3;19(1):216. doi: 10.1186/s12883-019-1445-9. PMID 31481010

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03924791/Prot_SAP_001.pdf